CLINICAL TRIAL: NCT06917690
Title: Multi-centeR, Open-label Study to EValuate the Safety, Efficacy, and Pharmacokinetics of FIlsuVEz (Oleogel-S10) in Japanese Subjects With Epidermolysis Bullosa (REVIVE)
Brief Title: A Study to Learn About the Safety and Efficacy of the Drug Oleogel-S10 in Japanese Patients With Epidermolysis Bullosa
Acronym: REVIVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-FILSVAA2-01
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Epidermolysis Bullosa; Junctional Epidermolysis Bullosa; Epidermolysis Bullosa, Dystrophic; Epidermolysis Bullosa, Junctional; Skin Abnormalities; Connective Tissue Disease; Collagen Diseases; Skin Diseases; Genetic Diseases, Inborn; Congenital Abnormalities
Keywords: Filsuvez; Birch Bark extract
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica; Skin Abnormalities; Connective Tissue Diseases; Collagen Diseases; Skin Diseases; Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oleogel-S10 (Experimental)
  Interventions: Drug: Oleogel-S10

INTERVENTIONS:
Drug: Oleogel-S10 — Topical gel

SUMMARY:
The goal of this clinical trial is to learn if Oleogel-S10 gel works to treat skin wounds from two types of inherited epidermolysis bullosa (EB): junctional EB (JEB) or dystrophic EB (DEB) in the Japanese population. Children and adults may participate. The trial also looks at the safety of Oleogel-S10 gel. The main questions it will answer are:

* Does Oleogel-S10 gel close wounds from JEB or DEB within 45 days or reduce the size of the wounds?
* Are there any medical problems when using Oleogel-S10 gel?
* How much of the drug ends up in your blood?

The study has 2 parts. In Part 1, participants will:

* Apply Oleogel-S10 gel to the EB wound dressings at least once every 4 days for 45 days.
* Visit the clinic once every 2 weeks for checkups and tests. If participants complete Part 1, they may participate in Part 2 if they choose to. In Part 2, participants will continue to receive Oleogel-S10 gel until the product is available to buy in Japan or until the trial is stopped by the company.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 21 days
2. Confirmed diagnosis of either JEB or DEB
3. Both biological parents and all 4 grandparents of Japanese descent
4. At least 3 EB wounds that meet the following criteria at the time of enrollment:

   * All are located outside of the anogenital region
   * All are distinguishable from any other wounds on the subject's body (separated by a minimum of 5 cm)
   * At least one has been present for a minimum of 21 days but less than 9 months AND is 10 cm2 to 50 cm2 in size
   * At least two have been present for a minimum of 21 days but less than 9 months AND/OR are 10 cm2 to 50 cm2 in size
5. A female subject must meet one of the following criteria:

   * If of childbearing potential, she must:

     1. Have a negative pregnancy test result at Screening and Baseline Visits, AND
     2. Agree to use one of the following highly reliable methods of contraception from the day of the informed consent signature until the day after the last Oleogel- S10 application. The following methods are acceptable:

        * Placement of an intrauterine device (IUD) or intrauterine releasing system (IUS)
        * Combined (both estrogen and progestogen) hormonal contraception (oral) associated with inhibition of ovulation, supplemented with a barrier method (preferably male condom)
        * Bilateral tubal occlusion
        * Sexual abstinence, defined as refraining from heterosexual intercourse during the entire study period
        * Partner vasectomy, provided that the partner is the sole sexual partner and has received medical verification of the surgical success
   * Be of non-childbearing potential, defined as one of the following:

     * Pre-menarche, OR
     * Post-menopausal (12 consecutive months of amenorrhea without an alternative medical cause), OR
     * Permanently sterile following hysterectomy, bilateral salpingectomy, or bilateral oophorectomy (supporting evidence required)
6. Subject and/or subject's legal representative has been informed about the study, has read and understood the information provided, and has given written informed consent
7. Subject and/or subject's legal representative is able and willing to follow all study procedures and instructions

Exclusion Criteria:

1. Hypersensitivity to Oleogel-S10 or any of its excipients
2. Diagnosis of EB subtypes simplex or Kindler EB
3. Receipt of systemic antibiotics for wound-related infections within 7 days prior to enrollment
4. Receipt of systemic or topical (on EB wounds) steroids within 30 days prior to enrollment Exceptions: Inhaled, ophthalmic, or mucosal applications, such as budesonide suspension for esophageal strictures
5. Receipt of immunosuppressive therapy or cytotoxic chemotherapy within 60 days prior to enrollment Note: Dupilumab to manage pruritis is allowed if the subject has been on a stable dose for more than 3 months prior to baseline
6. Receipt of systemic gene therapy for the treatment of inherited EB
7. Receipt of short-acting stem cell therapy (infusion of Muse cells, allogeneic adipocyte-derived MSC sheet (topically applied), TEMCELL (allogeneic MSCs, subcutaneous injection)) within 6 months prior to study enrollment
8. Receipt of topical gene therapy for the treatment of inherited EB (e.g., beremagene geperpavec) within 3 months prior to enrollment
9. Receipt of a JACE® skin graft on any of the target wounds
10. Current and/or former malignancy, including skin malignancies such as basal cell carcinoma and squamous cell carcinoma
11. Females: Pregnant or lactating, or of childbearing potential with a fertile male partner and unwilling to use a highly reliable method of contraception from the informed consent signature until study participation ends
12. Enrollment in any other interventional study or treated with any other investigational drug for any disease within 4 weeks prior to enrollment
13. Presence of any factor in the subject and/or legal representative that could interfere with study compliance, such as the ability to attend the scheduled study visits or to properly manage the dressing changes at home

Min Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Oleogel-S10 in Part I | Enrollment to 45 days
  The number and percentage of closed wounds within Part I (up to Day 45).

SECONDARY OUTCOMES:
To continue to evaluate the efficacy of Oleogel-S10 up to Day 90 in Part II | Enrollment to 90 days
  Evaluations will include the proportion of participants achieving complete wound closure of at least one target wound, the change in surface area of the wound, patient and clinician impression of improvement, frequency of dressing changes, and incidence of wound infections.
To evaluate the safety and tolerability of Oleogel-S10 in Part I and Part II | Enrollment through study completion, which is estimated for 2029
  Safety will be assessed through monitoring of adverse events, physical examinations, clinical laboratory tests (blood and urine samples), and vital signs from baseline up to study completion.
To evaluate the extent of systemic exposure to betulin | Enrollment to 45 days
  The concentration of betulin in blood at baseline and on Day 45.

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Fukuoka Children's Hospital - Dermatology, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Kobe University Hospital, Kobe
  - Niigata University Medical and Dental Hospital, Niigata
  - Toho University Omori Medical Center, Ōta-ku
  - Hokkaido University Hospital, Sapporo

IPD SHARING:
Plan to Share IPD: Yes